CLINICAL TRIAL: NCT01220947
Title: A Study of Danoprevir Boosted With Low Dose Ritonavir in Combination With Pegasys and Copegus in Treatment-Naive Patients With Chronic Hepatitis C Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NV22776; 2010-019584-10
Record Dates: First submitted 2010-10-07; First posted 2010-10-14 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; danoprevir; peginterferon alfa-2a; Ritonavir

ARMS (5):
- Group A (Experimental): Danoprevir 200 mg twice a day (BID) + ritonavir 100 mg + Pegasys 180 microgram sc qw + Copegus 1000 mg or 1200 mg po daily for 24 weeks
  Interventions: Drug: Copegus; Drug: Danoprevir; Drug: Pegasys; Drug: Ritonavir
- Group B (Experimental): Danoprevir 100 mg BID + ritonavir 100 mg + Pegasys 180 microgram sc qw + Copegus 1000 mg or 1200 mg po daily for 24 weeks
  Interventions: Drug: Copegus; Drug: Danoprevir; Drug: Pegasys; Drug: Ritonavir
- Group C (Experimental): Danoprevir 50 mg BID + ritonavir 100 mg + Pegasys 180 microgram sc qw + Copegus 1000 mg or 1200 mg po daily for 24 weeks
  Interventions: Drug: Copegus; Drug: Danoprevir; Drug: Pegasys; Drug: Ritonavir
- Group D (Experimental): Danoprevir 100 mg BID + ritonavir 100 mg + Pegasys 180 μg sc qw + Copegus 1000 mg or 1200 mg po daily for 12 weeks or 24 weeks
  Interventions: Drug: Copegus; Drug: Danoprevir; Drug: Pegasys; Drug: Ritonavir
- Group E (Active Comparator): Pegasys 180 microgram sc qw + Copegus 1000 mg or 1200 mg po daily for 48 weeks
  Interventions: Drug: Copegus; Drug: Pegasys

INTERVENTIONS:
Drug: Copegus — Copegus 1000 mg or 1200 mg po daily for 24 weeks.
Drug: Danoprevir — Danoprevir 50 mg BID
  Arms: Group C
Drug: Danoprevir — Danoprevir 100 mg BID
  Arms: Group B; Group D
Drug: Danoprevir — Danoprevir 200 mg BID
  Arms: Group A
Drug: Pegasys — Pegasys 180 microgram sc qw
Drug: Ritonavir — Ritonavir 100 mg
  Arms: Group A; Group B; Group C; Group D

SUMMARY:
This randomized, open-label, active-controlled, parallel-group study will evaluate the sustained virological response of danoprevir boosted with low dose ritonavir in combination with Pegasys (peginterferon alfa-2a) and Copegus versus Pegasys and Copegus alone in treatment-naive patients with chronic Hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients, >/=18 years of age
* Chronic Hepatitis C, Genotype 1 and 4
* HCV RNA >/=50,000 IU/mL
* treatment-naive

Exclusion Criteria:

* Patients with cirrhosis or incomplete/transition to cirrhosis
* Patients with other forms of liver disease, HIV infection, hepatocellular carcinoma or severe cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Sustained virological response (HCV RNA measured by Roche COBAS TaqMan HCV test) | 24 weeks after end of treatment

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | from baseline up to 72 weeks
Evaluation of relapse rate | up to 24 weeks after end of treatment
Characterization of resistance profile (HCV RNA sequencing and/or phenotypic analyses) | from baseline up to 72 weeks
Virological response at scheduled visits over time (HCV RNA measured by Roche COBAS TaqMan HCV test) | From baseline up to 72 weeks
Evaluation of virological breakthrough (viral load rebound) rate | up to 72 weeks
Evaluation of pharmacokinetics (serum concentrations assessed by validated methods) | up to 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (61):
- United States (23):
  - La Jolla, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Orlando, Florida
  - South Miami, Florida
  - Decatur, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Lutherville, Maryland
  - Detroit, Michigan
  - Manhasset, New York
  - New York, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Fayetteville, North Carolina
  - Medford, Oregon
  - Providence, Rhode Island
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Newport News, Virginia
- Vienna, Austria
- Brazil (3):
  - Salvador, Estado de Bahia
  - Porto Alegre, Rio Grande do Sul
  - Ribeirão Preto, São Paulo
- Canada (6):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Ottawa, Ontario
  - Toronto, Ontario
- France (7):
  - Clichy
  - Créteil
  - Marseille
  - Paris
  - Rennes
  - Toulouse
  - Vandœuvre-lès-Nancy
- Germany (6):
  - Berlin
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Hamburg
  - Leipzig
  - Würzburg
- Italy (6):
  - Bari, Apulia
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Milan, Lombardy
  - Pavia, Lombardy
  - Novara, Piedmont
- Mexico (2):
  - Guadalajara
  - Monterrey
- Santurce, Puerto Rico
- Spain (4):
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Seville, Sevilla
- United Kingdom (2):
  - London
  - Nottingham